CLINICAL TRIAL: NCT03524989
Title: The Effect of Hyperbaric Oxygen Therapy on Aerobic and Anaerobic Physical Fitness
Acronym: SPORTRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, MD, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0244-16-ASF
Record Dates: First submitted 2018-04-30; First posted 2018-05-15 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Healthy; Athletes
Keywords: hbot; hyperbaric oxygen; sport; mitochondria; athletes; aerobic
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized blinded controlled 2 groups with SHAM treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Hyperbaric Oxygen Therapy: 2 months of treatment consisting of 40 daily sessions, 60 minutes of 100% oxygen at pressure of 2 ATA each, five days a week
  Interventions: Device: Hyperbaric Oxygen Therapy
- Control/Crossover (Sham Comparator): SHAM therapy: 2 months of treatment consisting of 40 daily sessions, 60 minutes of 21% oxygen at pressure of 1.01 ATA each, five days a week
  Interventions: Device: SHAM treatment

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — 40 daily sessions, 60 minutes of 100% oxygen at pressure of 2 ATA each, five days a week for 2 months.
  Arms: Treatment
Device: SHAM treatment — 40 daily sessions, 60 minutes of 21% oxygen at pressure of 1.01 ATA each, five days a week for 2 months.
  Arms: Control/Crossover

SUMMARY:
Previous evidence showed hyperbaric oxygen can enhance aerobic and anaerobic performance during the exposure. The effect of continuous exposure of hyperbaric oxygen on performance was never evaluated.

DETAILED DESCRIPTION:
In recent years, several options for physical performance enhancement by increasing blood oxygen content were explored. One option is increasing the number of red blood cells by blood transfusions. Another option is using the erythropoietin hormone. These methods showed an effective increase of maximal oxygen consumption rate (VO2MAX) by 10%. However, due to their inherent risks, the international sports associations banned their uses. A third option of training in high altitude environments, but this option was never proved to be effective.

Another strategy would be increasing the blood oxygen content by increasing the plasma dissolved oxygen concentration. This would only be possible using hyperbaric oxygen therapy -which includes inhaling 100% oxygen in a pressure higher than the normal atmospheric pressure.

Previous evidence showed hyperbaric oxygen can enhance aerobic and anaerobic performance during the exposure. These studies evaluated the effect during a single hyperbaric oxygen exposure. The effect of continuous exposure of hyperbaric oxygen on performance was never evaluated.

The study is designed as a randomized controlled study aiming to evaluate the therapeutic effects of hyperbaric oxygen therapy (HBOT) on the aerobic and anaerobic performance.

After signing an informed consent form, patients will be randomized into 2 groups: treatment and control group. Patients will be invited for baseline evaluations. All patients would be evaluated 2 times - at baseline and after 2 months of follow up, The evaluation will include physical examination, VO2MAX, muscle biopsy for mitochondrial function, aerobic function measurements, cognitive assessment, brain MRI, brain EEG.

Protocols:

Treatment: Patients will receive 40 daily sessions, 5 days/week, 60 minutes each with 5 minutes air break every 30 minutes, 100% oxygen at 2 atmospheres (ATA).

Control: Patients will receive 40 daily sessions, 5 days/week, 60 minutes each with 5 minutes air break every 30 minutes, 21% oxygen (air) at 1.01 ATA.

Upon completion of the study, control group would be offered to crossover and complete additional 40 sessions of 100% oxygen at 2 ATA. A third evaluation would be performed in case patients will complete the protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 or 40-50 age
* Professional performance of aerobic sports for ages 18-25 (at least 5 times a week)
* Moderate and above performance of aerobic sports for ages 40-50 (at least 4 times a week)
* no chronic illness
* no significant musculoskeletal injury in the past 3 months

Exclusion Criteria:

* Debilitating significant musculoskeletal injury
* Previous hyperbaric oxygen exposure
* Lung pathology
* Middle or Inner ear pathology
* Claustrophobia
* Chronic illness
* Smoking
* Chronic medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline of exercise VO2 MAX at 2 months and 4 months | baseline, at 2 months, 4 months
  Using a standard exercise test which includes gas analysis, the change in VO2 maxs will be assessed 2 months and 4 months compared to baseline

SECONDARY OUTCOMES:
Change from baseline of maximal respiratory rate | baseline, at 2 months, at 4 months
  Using a trucut needle, the gluteus maximus will be sampled in a sterile technique for 1-2mg of muscle tissue. Oroboros O2k high resolution respirometry analyzer will be used (Oxygraph-2k Oroboros Instruments, Innsbruck, Austria). Maximal respiration rate (nmol/ml) will be calculated.
Change from baseline of basal respiration rate | baseline, at 2 months, at 4 months
  Using a trucut needle, the gluteus maximus will be sampled in a sterile technique for 1-2mg of muscle tissue. Oroboros O2k high resolution respirometry analyzer will be used (Oxygraph-2k Oroboros Instruments, Innsbruck, Austria). Basal respiration rate (nmol/ml) will be measured where mitochondrial reserve capacity and ATP-linked respiration will be calculated.
Change from baseline of respiration independent adenosine triphosphate (ATP) production (in muscle biopsy | baseline, at 2 months, at 4 months
  Using a trucut needle, the gluteus maximus will be sampled in a sterile technique for 1-2mg of muscle tissue. Oroboros O2k high resolution respirometry analyzer will be used (Oxygraph-2k Oroboros Instruments, Innsbruck, Austria). Inpendent adenosine triphosphate (ATP) production (proton leak) (nmol/ml) will be calculated.
Change from baseline in body fat/muscle ratio | baseline, at 2 months, at 4 months
  Using an electric current weight, the fat % and muscle % content will be measured.
Change in maximal vertical jump (meters) | baseline, at 2 months, at 4 months
  Maximal running speed, maximal vertical jump height will be measured according the standards.
Change in maximal running speed (km/hr) | baseline, at 2 months, at 4 months
  Maximal running speed will be measured according the standards.
Change in forced expiratory volume at one second (FEV1) | baseline, at 2 months, at 4 months
  Using a standard spirometry, forced expiratory volume at one second (FEV1) (liters/second) will be measured
Change in forced volume capacity (FVC) | baseline, at 2 months, at 4 months
  Using a standard spirometry, forced volume capacity (FVC) (liters/second) will be measured
Change in general cognitive function | baseline, at 2 months, at 4 months
  Patients' cognitive functions will be assessed by Neurotrax computerized cognitive tests to generate the general cognitive index (0-100)
Change from baseline of brain blood perfusion in brain MRI | baseline, at 2 months, at 4 months
  imaging will be performed for evaluation of brain changes and angiogenesis process using MRI perfusion and microstructure

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ramla, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hadanny A, Hachmo Y, Rozali D, Catalogna M, Yaakobi E, Sova M, Gattegno H, Abu Hamed R, Lang E, Polak N, Friedman M, Finci S, Zemel Y, Bechor Y, Gal N, Efrati S. Effects of Hyperbaric Oxygen Therapy on Mitochondrial Respiration and Physical Performance in Middle-Aged Athletes: A Blinded, Randomized Controlled Trial. Sports Med Open. 2022 Feb 8;8(1):22. doi: 10.1186/s40798-021-00403-w. PMID 35133516